CLINICAL TRIAL: NCT02831465
Title: Dynamic Hyperinflation During Maximal Voluntary Ventilation in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B076201318918
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-07

CONDITIONS: Dynamic Hyperinflation
Keywords: Dynamic hyperinflation; Maximal Voluntary Ventilation; Inspiratory capacity; healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy subjects (Experimental): Subjects with normal lung function between 40 and 70 years old.
  Interventions: Behavioral: Healthy Subjects

INTERVENTIONS:
Behavioral: Healthy Subjects — Subjects with normal lung function performed MVV at increasing breathing frequencies and maximal tidal volume, from 10 to 100 cycles per minute. Inspiratory capacity (IC) was measured at rest and after each 12 seconds of MVV in order to detect DH. From the moment DH appeared at a given frequency, only one additional MVV at a higher breathing frequency was conducted to confirm DH.

SUMMARY:
Maximal Voluntary Ventilation (MVV) correlates well with maximal exercise capacity and is used to assess the ventilatory function during exercise in COPD (Chronic Obstructive Pulmonary Disease) patients. Dynamic hyperinflation (DH) often occurs during MVV in COPD and is believed to be due to expiratory flow limitation.

The present study is intended to assess whether DH can also occur during MVV in normal subjects without expiratory flow limitation.

DETAILED DESCRIPTION:
Maximal voluntary ventilation (MVV) correlates well with maximal exercise capacity and is used to assess the ventilatory function during exercise in COPD (Chronic Obstructive Pulmonary Disease) patients. Dynamic hyperinflation (DH) often occurs during MVV in COPD and is believed to be due to expiratory flow limitation. The present study is intended to assess whether DH can also occur during MVV in normal subjects without expiratory flow limitation.

Study design: healthy subjects with normal lung function will perform MVV at increasing breathing frequencies and maximal tidal volume, from 10 to 100 cycles per minute. Inspiratory capacity (IC) will be measured at rest and after each 12 seconds of MVV in order to detect DH. From the moment DH appeares at a given frequency, only one additional MVV at a higher breathing frequency will be conducted to confirm DH.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* History of asthma, obstructive syndrome on basic lung function

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Frequency which induces Dynamic Hyperinflation | day one
  We analyze Frequency of Maximal Voluntary Ventilation (MVV) which induces a significant decrease of the Inspiratory Capacity (IC) post MVV compared to the IC at rest.

SECONDARY OUTCOMES:
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and Forced Expiratory Volume in one second | day one
  We analyze if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and Forced Expiratory Volume in one second
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and Forced Vital Capacity | day one
  We analyze if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and Forced Vital Capacity
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and Forced Expiratory Flows at 25%, 50% and 75% of Forced Vital Capacity | day one
  We analyze if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and Forced Expiratory Flows at 25%, 50% and 75% of Forced Vital Capacity
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and age | day one
  We analyze if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and age
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and body mass index | day one
  We analyze if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and body mass index
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and Inspiratory Capacity at rest | day one
  We analyzed if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and Inspiratory capacity at rest
Correlation between the frequency which induces Dynamic Hyperinflation (DH) and IC/FVC ratio (IC : Inspiratory Capacity at rest ; FVC : Forced Vital Capacity) | day one
  We analyze if there is a good correlation between the frequency which induces a significant Dynamic Hyperinflation (DH) and IC/FVC ratio (IC : Inspiratory Capacity at rest ; FVC : Forced Vital Capacity)
Comparison Maximal Voluntary Ventilation with Forced Expiratory Volume in one second multiplied by 35 | day one
  We compare Maximal Voluntary Ventilation at the different frequencies with the common predictive value of maximal ventilation obtained by multiplying Forced Expiratory Volume in one second by 35

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ninane, MD, PhD, Principal Investigator — University Hospital Center Saint Pierre chest service
Locations (1):
- CHU St. Pierre, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No